CLINICAL TRIAL: NCT06501079
Title: The Efficacy of Dexamethasone Versus Magnesium Sulphate Added to Bupivacaine Used in Erector Spinae Plane Block for Perioperative Pain Control in Patients Undergoing Unilateral Nephrectomy
Brief Title: Dexamethasone Versus Mg Added to Bupivacaine Used in ESPB for Perioperative Pain Control in Patients Undergoing Unilateral Nephrectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Soliman, lecturer of anesthesia, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AP2404-201-004
Record Dates: First submitted 2024-06-29; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Renal Neoplasm
Keywords: Dexamethasone; Magnesium Sulphate; Bupivacaine; Erector Spinae Plane Block; perioperative; pain control; unilateral nephrectomy
MeSH Terms: conditions — Kidney Neoplasms; Agnosia

STUDY DESIGN:
Intervention Model Description: The aim of the current study is to compare the effect of adding dexamethasone versus magnesium sulphate to bupivacaine in ultrasound-guided erector spinae plane block on the severity of postoperative pain.
  Primary Objectives to compare the effect of ESPB without additives to the effect of adding dexamethasone and to the effect of adding magnesium sulphate in the form of post-operative visual analogue scale (VAS) after 30 hours at rest.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Normal saline (Active Comparator): receiving erector spinae block with 27ml bupivacaine 0.25% + 3 ml NS
  Interventions: Procedure: ultrasound guided Erector Spinae Plane Block using 27ml bupivacaine 0.25%
- magnesium sulphate 10% (Active Comparator): receiving erector spinae block with 27 ml bupivacaine 0.25% + 3 ml magnesium sulphate 10%
  Interventions: Procedure: ultrasound guided Erector Spinae Plane Block using 27ml bupivacaine 0.25%
- dexamethasone (Active Comparator): receiving erector spinae block with 27 ml bupivacaine 0.25% + 8 mg dexamethasone (2 ml) + 1 ml NS.
  Interventions: Procedure: ultrasound guided Erector Spinae Plane Block using 27ml bupivacaine 0.25%

INTERVENTIONS:
Procedure: ultrasound guided Erector Spinae Plane Block using 27ml bupivacaine 0.25% — ESP block will be performed U/S at the level of T 10 paraspinal level. The ultrasound transducer should be placed in the midline of the back at the desired level. The probe should then slowly be moved laterally until the transverse process is visible. The transverse process requires differentiation from the rib at that level.
  Erector spinae muscle should be identified superficial to the transverse process. The needle inserted superior to the ultrasound probe in the cephalad to caudal direction. Once the needle tip is below the erector spinae muscle.
  This separation from the transverse process confirms the proper needlemposition.
  The local anesthetic should then be injected in 5 ml increments. The block will be performed preoperatively.

SUMMARY:
Aim of the study:

The current study aims to compare the effect of adding dexamethasone versus magnesium sulfate to bupivacaine in ultrasound-guided erector spinae plane block on the severity of postoperative pain.

Primary Objectives:

- To compare the effect of ESPB without additives to the effect of adding dexamethasone and to the impact of adding magnesium sulfate in the form of post-operative morphine consumption

DETAILED DESCRIPTION:
Aim of the study:

The current study aims to compare the effect of adding dexamethasone versus magnesium sulfate to bupivacaine in ultrasound-guided erector spinae plane block on the severity of postoperative pain and postoperative morphine consumption.

Methodology:

I. Study design:

This is a randomized Controlled Study. It will involve three groups: Control Group (C) receiving erector spinae block with 27ml bupivacaine 0.25% + 3 ml NS, Group (M) receiving 27 ml bupivacaine 0.25% + 3 ml magnesium sulphate 10%, Group (D) receiving 27 ml bupivacaine 0.25% + 8 mg dexamethasone (2 ml) + 1 ml NS.

II. Study setting and location:

National Cancer Institute, Cairo University after approval by the institutional review board.

III. Study population:

Adult patients undergoing unilateral nephrectomy under general anesthesia.

Patients will be randomly assigned to the groups using online random number generator.

Erector Spinae Plane Block technique:

Informed consent, including the risks and benefits of the procedure, should be obtained before carrying out an ESP block. A peri-procedural "timeout" should be performed to confirm the type, side, and location of the procedure and ensure that there are no contraindications.

Standard patient monitoring should be in place, including continuous ECG monitoring, pulse oximetry, and blood pressure measurement in at least 5-minute intervals. Patients should be prepped and draped in sterile conditions. Sterile gloves and surgical cap and a mask are necessary, and the ultrasound probe is placed into the sterile ultrasound probe cover for imaging. The ESP block will be performed at the level of T 10 paraspinal level. The ultrasound transducer should be placed in a cephalocaudal orientation over the midline of the back at the desired level. The probe should then slowly be moved laterally until the transverse process is visible. The transverse process requires differentiation from the rib at that level. The transverse process will be more superficial and wider, while the rib will be deeper and thinner. Erector spinae muscle should be identified superficial to the transverse process. The needle should be inserted superior to the ultrasound probe using an in-plane approach in the cephalad to caudal direction. Once the needle tip is below the erector spinae muscle, a small bolus of local anesthetic should be given through the needle. The erector spinae muscle should be visualized, separating from the transverse process. This separation from the transverse process confirms the proper needle position.

The local anesthetic should then be injected in 5 ml increments, with aspiration after every 5 ml to prevent intravascular injection. Block will be performed preoperatively in the preoperative holding area.

Heart rate and blood pressure to be recorded preoperative, intraoperative and postoperatively

Assessment of pain:

Pain assessment will be done through Visual Analogue Scale. Patients should be informed preoperatively about it and how to use this scale. Starting from recovery time, pain assessment is done by asking the patient to mark the intensity of pain perceived and express it on a 10 cm horizontal scale ranging from no pain at one end to the worst possible pain at the other end.

Assessment of pain is to be done in the recovery unit and at 0,2,4,8,12,18, 24 and 30 hours postoperatively.

Total amount of opioid needed in first 24 hours to be recorded.

Rescue Analgesia:

Intraoperative rescue analgesia will be done by giving fentanyl at dose of 1 mic/Kg. Postoperatively, NSAIDs such as Ketorolac 30 mg I.V infusion if VAS is between 3 to 6, and Morphine 3 mg I.V if VAS equals or is more significant than 6.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 - 65)
* Patients undergoing unilateral nephrectomy
* ASA II / III

Exclusion Criteria:

* Patient refusal
* Age less than 18 years
* Allergy to any of the studied medications
* Mid line incision
* Bilateral nephrectomy
* Distorted anatomy of the back (e.g. kyphoscoliosis)
* Known neurologic disorders, psychiatric disorder or chronic pain
* Local infection
* Hemodynamic instability

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
postoperative opioid consumption | 24 hours post-operatively
  total postoperative rescue analgesia be by Morphine

SECONDARY OUTCOMES:
time of first rescue analgesia | during 1st 24 postoperatively.
  Ketorolac 30 mg I.V infusion if VAS is between 3 to 6, and Morphine 3 mg I.V if VAS equals or greater than 6
Intraoperative opioid consumption | intraoperative
  total Intraoperative rescue analgesia will be done by giving fentanyl at dose of 1 mic/Kg
visual analogue scale 30 hours post-operatively at rest | 24 hours post-operatively at rest
  visual analogue scale from 0 to 10 as 0 no pain and 10 worst pain

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer institute - Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Till publication